CLINICAL TRIAL: NCT00003709
Title: Phase I and Pharmacokinetic Study of FB-642 Administered Orally on a Weekly Schedule to Patients With Advanced Solid Tumors
Brief Title: Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Therapy and Research Center, Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066817; P30CA054174 (NIH); UTHSC-9895011080 (Other: UTHSCSA IRB); ILEX-FB-642-101 (Other: Proctor and Gamble); SACI-IDD-98-21 (Other: San Antonio Cancer Institute); NCI-V98-1503 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-08-17 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — carbendazim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carbendazim — Patients receive oral carbendazim weekly for 3 weeks followed by 1 week of rest. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxic effects. Cohorts of 3-6 patients receive escalating doses of carbendazim. If dose limiting toxicity (DLT) is seen in 1 of 3 patients treated at a given dose level, 3 additional patients will be entered at the same dose level. Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT. Patients are followed for up to 30 days posttreatment.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of carbendazim in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oral carbendazim in patients with advanced solid tumors. II. Determine the qualitative and quantitative toxic effects of oral carbendazim in these patients. III. Characterize the pharmacokinetic profile of oral carbendazim in these patients. IV. Assess the recommended dose of oral carbendazim to be used in phase II studies. V. Determine preliminary evidence of antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral carbendazim weekly for 3 weeks followed by 1 week of rest. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxic effects. Cohorts of 3-6 patients receive escalating doses of carbendazim. If dose limiting toxicity (DLT) is seen in 1 of 3 patients treated at a given dose level, 3 additional patients will be entered at the same dose level. Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT. Patients are followed for up to 30 days posttreatment.

PROJECTED ACCRUAL: Up to 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically proven advanced solid tumors for which no standard therapy exists or that has progressed or recurred following prior therapy Measurable or evaluable disease No hematological malignancies (e.g., leukemia or lymphoma) No known brain or leptomeningeal disease, unless lesions were previously irradiated, currently not being treated with corticosteroids, and have no clinical symptoms

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin less than 1.5 mg/dL AST or ALT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if due to tumor) PT and aPTT no greater than 1.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No unstable atrial or ventricular arrhythmias that require medication No ischemic events within 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No psychiatric disorders No history of seizure disorders No other severe concurrent disease No history of ulcers or abnormalities that would interfere with carbendazim absorption No history of hypersensitivity to PEG-formulated medications (including cyclosporine or etoposide)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas or mitomycin) and recovered No concurrent cytotoxic therapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: No prior gastrointestinal surgery that would interfere with carbendazim absorption Other: No concurrent use of phenytoin, phenobarbital, valproic acid, or other antiepileptic prophylaxis No concurrent scheduled antacids, such as H2 blockers (e.g., cimetidine or ranitidine) or hydrogen pump inhibitors (e.g., omeprazole), or cisapride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-10; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, MD, Study Chair — San Antonio Cancer Institute
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas